CLINICAL TRIAL: NCT02637869
Title: Evaluating Community Health Centers' Adoption of a New Global Capitation Payment
Acronym: eCHANGE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: OCHIN, Inc. (Other); Robert Wood Johnson Foundation (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Heintzman, Principal Investigator, Oregon Health and Science University
Other Study IDs: AHRQ R01HS22651; 71125 (Other Grant/Funding Number: AHRQ)
Record Dates: First submitted 2015-12-02; First posted 2015-12-22 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Chronic Diseases
Keywords: Health Expenditures; Prospective Payment System; Health Care Utilization; Health Care Quality, Access, and Evaluation
MeSH Terms: conditions — Chronic Disease; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group - non-intervention: Clinics that did not participate in the APM project
- Alternative Payment Model -intervention: Oregon developed an Alternative Payment Methodology (APM). Under this APM pilot participating CHCs will receive a prospective payment system (PPS) payment as a capitated equivalent in a per-member-per-month rate for all of their Medicaid patients
  Interventions: Other: Alternative Payment Model

INTERVENTIONS:
Other: Alternative Payment Model — Oregon developed an Alternative Payment Methodology (APM). Under this APM pilot participating CHCs will receive a prospective payment system (PPS) payment as a capitated equivalent in a per-member-per-month rate for all of their Medicaid patients
  Groups: Alternative Payment Model -intervention

SUMMARY:
The investigators are conducting a prospective analysis of the Alternative Payment Methodology (APM) demonstration project sites. The investigators' goal is to conduct a cross project analysis of findings. The investigators propose to use mixed methods to study processes and outcomes associated with the APM natural experiment in payment reform. The investigators hypothesize that Community Health Centers (CHCs) participating in the APM demonstration project will redesign their workflows to better focus on patient and population health needs, resulting in reallocation of financial resources, lower overall costs, changes in utilization patterns, and improved quality.

DETAILED DESCRIPTION:
Led by the Oregon Primary Care Association, three community health center (CHC) organizations in Oregon developed an Alternative Payment Methodology (APM). Under this APM pilot participating CHCs will receive a prospective payment system (PPS) payment as a capitated equivalent in a per-member-per-month rate for all of their Medicaid patients. Oregon CHC organizations (several clinic sites) implemented Phase I of this demonstration project on March 1, 2013; Phase II A was implemented on July 1, 2014; Phase II B on October 1, 2014; and Phase III began July 1, 2015.

We are a prospective analysis of the APM project sites. We propose to use mixed methods to study processes and outcomes associated with the APM natural experiment in payment reform. We hypothesize that CHCs participating in the APM demonstration project will redesign their workflows to better focus on patient and population health needs, resulting in reallocation of financial resources, lower overall costs, changes in utilization patterns, and improved quality.

The study will include baseline qualitative data collection as clinics are transitioning to the APM methodology. We will conduct 2 site visits to each intervention clinic to observe practice changes that occurred post APM-implementation (first visit approximately 12-18 months post-APM implementation; second visit approximately 30-36 months post-APM implementation). We will also assemble and analyze of pre-post quantitative and qualitative datasets, and interpretation and dissemination of study findings.

ELIGIBILITY:
Inclusion Criteria:

1. Total clinic population:

   established patients at intervention and control clinics aged 2-64
2. Medicaid Population:

Medicaid-enrolled patients at intervention and control clinics aged 2-64

Exclusion Criteria:

1. Total clinic population:

   non-established patients at intervention and control clinics aged 2-64
2. Medicaid Population:

non-Medicaid-enrolled patients at intervention and control clinics aged 2-64

Ages: 2 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community Health Center (CHC) and clinic patients of which CHCs are participating in the APM demonstration (intervention) or are matched with APM CHCs (control)
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Internal services utilization | ≤3 years pre-APM implementation and ≤3 years post
  Number and type of internal services utilized including number and ratio of "traditional" face to face visits vs. "nontraditional" encounters and communication via phone, personal health record, and email

SECONDARY OUTCOMES:
Quality care measures | ≤3 years pre-APM implementation and ≤3 years post
  We selected measures that are: 1) identified by Oregon's Medicaid program and/or those on the list of Clinical Quality Measures in the electronic health record (EHR) incentive programs; 2) feasibly measured with EHR or Medicaid claims data; 3) representative across age groups and gender; 4) representative of treatment levels (e.g., prevention, acute and chronic condition care); and 5) relevant to CHC populations.
External services utilization | ≤3 years pre-APM implementation and ≤3 years post
  Number and type of external services utilized including percent of patients with a follow-up appointment after discharge and average wait time
Medicaid expenditures | ≤3 years pre-APM implementation and ≤3 years post
  We will calculate the average pre-post APM difference in total Medicaid expenditures attributable to the subpopulation of Medicaid-insured patients in APM intervention clinics, subtracted by the average difference among Medicaid-insured patients in comparison clinics

OTHER OUTCOMES:
Study the change processes associated with APM implementation | ≤3 years pre-APM implementation and ≤3 years post
  Qualitative assessment of practice change through interviews and site visits

CONTACTS AND LOCATIONS:
Overall Officials: John Heintzman, MD, MPH, Principal Investigator — Oregon Health and Science University; Heather Angier, MPH, Study Director — Oregon Health and Science University

REFERENCES:
- [Background] Heintzman J, Cottrell E, Angier H, O'Malley J, Bailey S, Jacob L, DeVoe J, Ukhanova M, Thayer E, Marino M. Impact of Alternative Payment Methodology on Primary Care Visits and Scheduling. J Am Board Fam Med. 2019 Jul-Aug;32(4):539-549. doi: 10.3122/jabfm.2019.04.180368. PMID 31300574
- [Result] Angier H, O'Malley JP, Marino M, McConnell KJ, Cottrell E, Jacob RL, Likumahuwa-Ackman S, Heintzman J, Huguet N, Bailey SR, DeVoe JE. Evaluating community health centers' adoption of a new global capitation payment (eCHANGE) study protocol. Contemp Clin Trials. 2017 Jan;52:35-38. doi: 10.1016/j.cct.2016.11.001. Epub 2016 Nov 9. PMID 27836506
- [Result] Cottrell EK, Hall JD, Kautz G, Angier H, Likumahuwa-Ackman S, Sisulak L, Keller S, Cameron DC, DeVoe JE, Cohen DJ. Reporting From the Front Lines: Implementing Oregon's Alternative Payment Methodology in Federally Qualified Health Centers. J Ambul Care Manage. 2017 Oct/Dec;40(4):339-346. doi: 10.1097/JAC.0000000000000198. PMID 28857887

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT02637869/Prot_SAP_000.pdf